CLINICAL TRIAL: NCT04395807
Title: Helmet Continuous Positive Airway Pressure Versus High-Flow Nasal Cannula in COVID-19: A Pragmatic Randomised Clinical Trial
Brief Title: Helmet CPAP Versus HFNC in COVID-19
Acronym: COVID HELMET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1. Few eligible patients at study start
  2. Patients received HFNC prior to intermediate care ward admission
  3. NIV was locally considered a step-up therapy to HFNC
  4. Full-face masks replaced the Helmet interface as local NIV standard
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVID HELMET
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: COVID; Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Helmet CPAP (Active Comparator): Helmet Continuous Positive Airway Pressure (CaStar hood for CPAP therapy by Starmed/Intersurgical) driven by high-flow blender (Bio-Med Devices).
  Interventions: Device: Helmet CPAP
- HFNC (Active Comparator): High-Flow Nasal Cannula (OptiflowTM nasal high-flow interface) driven by AIRVO 2 humidification system (Fisher and Paykel)
  Interventions: Device: HFNC

INTERVENTIONS:
Device: Helmet CPAP — Start-up air flow 40 L/min. Start-up PEEP 5 cmH2O. Max PEEP 20 cmH2O. Oxygen flow / FiO2% according to 92% SpO2 target. Titrations at physician's choice.
  Arms: Helmet CPAP
Device: HFNC — Start-up air flow 30 L/min. Max air flow 60 L/min. Oxygen flow / FiO2% according to 92% SpO2 target. Titrations at physician's choice.
  Arms: HFNC

SUMMARY:
We aim to investigate whether the use of Continuous Positive Airway Pressure using a Helmet device (Helmet CPAP) will increase the number of days alive and free of ventilator within 28 days compared to the use of a High Flow Nasal Cannula (HFNC) in patients admitted to Helsingborg Hospital, Sweden, suffering from COVID-19 and an acute hypoxic respiratory failure.

DETAILED DESCRIPTION:
A detailed description can be found in the study protocol published in Trials in Dec 2020:

Tverring, J., Åkesson, A. & Nielsen, N. Helmet continuous positive airway pressure versus high-flow nasal cannula in COVID-19: a pragmatic randomised clinical trial (COVID HELMET). Trials 21, 994 (2020). https://doi.org/10.1186/s13063-020-04863-5

ELIGIBILITY:
Inclusion Criteria (all of the following):

1. Age ≥ 18 years
2. Sars-Cov-2 found in the upper or lower respiratory tract by PCR during the current disease episode
3. Peripheral oxygen saturation (SpO2) < 92 % despite conventional low-flow oxygen therapy of at least 6 L /min for at least 15 min
4. A decision to initiate HFNC or Helmet CPAP by the attending ward physician
5. The patient has given written informed consent to participate.

Exclusion Criteria (any of the following):

1. Need for direct admission to the intensive care unit for mechanical ventilation
2. Unconsciousness or drowsiness
3. Pneumothorax
4. Carbon dioxide pressure (pCO2) > 6 kPa in venous blood gas (VBG)
5. Underlying chronic obstructive pulmonary disease stage III-IV
6. A decision not to participate
7. Inability to comprehend the study content and give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Ventilator-Free Days (VFD) | 28 days
  Number of days alive and free of mechanical ventilation within 28 days. Patients who die within 28 days will be counted as 0 VFD. Time in ventilator will be counted in hours and rounded to whole days.

SECONDARY OUTCOMES:
SpO2/FiO2-ratio | 1 hour after randomisation
  Peripheral oxygen saturation divided by fraction of inspired oxygen
Patient comfort | 24 hours after randomisation
  Visual scale (1-10)
Frequency of endotracheal intubation | 28 days
  Min 0, Max 1
Frequency of carbon dioxide rebreathing | 28 days
  Defined as pCO2 > 6 kPa in a venous blood gas. Min 0, Max ∞
Days alive within | 28 days and 180 days
  All-cause mortality. (180 days endpoint not in primary publication)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Tverring, MD, Principal Investigator — Lund University
Locations (1):
- Helsingborg's Hospital, Helsingborg, Region Skane, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tverring J, Akesson A, Nielsen N. Helmet continuous positive airway pressure versus high-flow nasal cannula in COVID-19: a pragmatic randomised clinical trial (COVID HELMET). Trials. 2020 Dec 3;21(1):994. doi: 10.1186/s13063-020-04863-5. PMID 33272319